CLINICAL TRIAL: NCT02734927
Title: Motivation and Executive Control in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-A00026-37
Record Dates: First submitted 2016-03-07; First posted 2016-04-12 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; motivation; executive control
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- schizophrenia group (Active Comparator): Schizophrenia patients suffering
  Interventions: Other: realization of computerized exercises
- control group (Sham Comparator): subjects showing no psychological or neurological disorder
  Interventions: Other: realization of computerized exercises

INTERVENTIONS:
Other: realization of computerized exercises

SUMMARY:
In order to control a behaviour, investigators need to realise goal directed actions and to priories some actions. This control is required in unusual situation. Appropriate actions are selected and coordinated according to context and aim.

Several studies try to draw a model of executive function. Recently, Koechlin has suggested a three levelled organisation to explain how the prefrontal cortex controls actions.

Contextual control is useful to answer appropriately with the immediate context. Episodic control allows selecting the action according to specific information given before. Sensorial control is the automatic response when a stimulus is presented.

Some diseases like schizophrenia are associated with neurological dysfunction in prefrontal cortex. Chambon and al (2008) have identified a dysfunction of contextual control in schizophrenia.

As the prefrontal cortex is involved in motivational process, it seems interesting to study potential links between executive function and motivation. A study from Kouneiher shows contextual and episodic activation of motivation in healthy population.

Investigators aim to study the way motivational process are recruited in schizophrenia.

DETAILED DESCRIPTION:
behavioral protocol. Letters (vowel and consonant; upper- or lower- case) are presented in several colours into successive blocks. Each block included a series of eight letters. Each colour required a specific task given by a fixed rule (contextual control) but for some colour, the rule changes sometimes (episodic control). Participants are informed that payoffs vary according to their own performance. A frame indicates essay with bonus reward. Moreover a dashed frame indicates a low-bonus reward and a solid frame means a high-bonus reward. Thus different blocks are designed: low-incentive block and high incentive block.

This reward increased from standard to bonus motivation in high-incentive block (contextual motivation) and from low to high according to the type of blocks (episodic motivation) Reaction time may be higher in bonus reward Patients with schizophrenia are not sensitive to contextual motivation, and therefore patients should behave differently than control in contextual motivation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years old
* schizophrenia
* french native speaker

Exclusion Criteria:

* Neurological disease
* Motor or visual deficit
* Somatic treatment with neurological impact
* Drug abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
reaction time | 24 hours
  reaction time is recorded when the subject press the key (subject should press a key function of the characteristics of the letter submitted)Reaction time should vary with the level of executive control (episodic, contextual, and motivation control (episodic or contextual motivation). Responses will be compared across patients and control.

CONTACTS AND LOCATIONS:
Locations (1):
- Professeur FRANCK Nicolas, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No